CLINICAL TRIAL: NCT02207114
Title: Southeastern Pennsylvania Adult and Pediatric Prevention Epicenter Network - Randomized Control Trial
Brief Title: Using Biomarkers to Optimize Antibiotic Strategies in Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 813623
Record Dates: First submitted 2014-02-03; First posted 2014-08-01 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Sepsis
Keywords: Sepsis; Systemic Inflammatory Response Syndrome (SIRS); Antibiotic use; Intensive Care Unit
MeSH Terms: conditions — Sepsis; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observational (No Intervention): 9 blood biomarkers (including C reactive protein and Procalcitonin) will be assessed across 3 days. Results will not be shared with the subject's medical team. At 3 days, the definitive diagnosis of infection will be determined using Center for Disease Control (CDC) criteria; this will serve as the gold standard for determining biomarker test characteristics. Additional data to collect: demographics, comorbidities, medication use (like antibiotics), lab cultures, x-rays, sepsis resolution, length of hospital stay, and ultimate outcome (i.e., discharge, death). Phase I will identify the biomarker(s) providing the greatest negative predictive value in identifying patients at very low likelihood bacterial infection.
- Biomarker Algorithm Intervention (Experimental): The Algorithm arm is equivalent to the intervention. Biomarker algorithm along with the patient's biomarker assay results will be given to clinical team to assist in deciding to continue antibiotics.
  The intervention will consist of using the biomarker identified as useful in Phase I to compile an algorithm along containing the patient's biomarker assay results and providing this as additional information for a clinical team consider using to assist in deciding to continue antibiotics. Biomarker algorithms may be different for adult versus pediatric patients, and across different types of ICUs.
  Interventions: Other: Biomarker Algorithm Intervention

INTERVENTIONS:
Other: Biomarker Algorithm Intervention — The intervention will consist of using the biomarker identified as useful in Phase I to compile an algorithm along containing the patient's biomarker assay results and providing this as additional information for a clinical team consider using to assist in deciding to continue antibiotics. Biomarker algorithms may be different for adult versus pediatric patients, and across different types of ICUs.
  Arms: Biomarker Algorithm Intervention

SUMMARY:
The proposed work will provide critical insights into the potential impact of a biomarker-based algorithm on reducing unnecessary antibiotic use in different adult and pediatric/neonatal ICU's. This proposal will also assess the costs (or savings) of a biomarker-based intervention. Overall, the results of this work will be critical in informing future strategies to eliminate unnecessary antibiotic use and curb the continued rise in antimicrobial resistance.

DETAILED DESCRIPTION:
The goal of this project is reduce unnecessary use of antibiotics in the ICU. The purpose of Phase I of the study is to identify the biomarker, or combination of biomarkers, that provides optimal test characteristics in identifying adults and children/neonates with presumed sepsis who have a very low likelihood of bacterial infection. Results of Phase I will result in development of a biomarker-based algorithm to inform need for antibiotic use in ICU patients. In Phase II, the impact of this biomarker-based algorithm on reducing antibiotic use in the ICU will be determined. Costs or savings associated with the algorithm will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. SIRS Criteria

   SIRS is considered to be present when patients have more than one of the following clinical findings:
   * body temperature >38°C or <36°C
   * heart rate >90 min-1
   * respiratory rate of >20 min-1 or a Paco2 of <32 mm Hg
   * and a white blood cell count of >12,000 cells µL-1 or <4,000 µL-1
2. new empiric antibiotic therapy is initiated, indicating the suspicion of infection. Accepted criteria for SIRS will be used for the Medical Intensive Care Unit and Surgical Intensive Care Unit populations, with appropriate age-specific vital signs definitions to help make the definitions relevant for the Pediatric Intensive Care Unit population.

Exclusion Criteria:

1. a code status of "do not resuscitate"
2. absence of initiation or expansion of antibiotic therapy despite meeting criteria for sepsis
3. presence of an immunocompromising condition.

An immunocompromising condition will be defined as one of the following:

* human immunodeficiency virus (HIV) infection with a t-helper cell (CD4) count <200 cell/mm3; 2) immunosuppressive therapy after organ transplantation
* neutropenia (<500 neutrophils/mm3)
* active chemotherapy within the 3 months preceding eligibility or
* diagnosis of cystic fibrosis.

These criteria all represent conditions in which antibiotic use is much less likely to be decreased regardless of the results of a biomarker and are consistent with exclusion criteria used in past studies of the impact of biomarkers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2012-01; Primary Completion 2016-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Duration of antibiotic therapy started upon enrollment for presumed sepsis | Two years
  The primary outcome is the duration of antibiotic treatment after enrollment, expressed in days. This variable will focus specifically on the antibiotic agents given for the episode of presumed sepsis for which the patient was included in the study.

SECONDARY OUTCOMES:
Subject's Final Disposition | Participants will be followed for the duration of hospital stay, an expected average of 6 days
  This includes assessing ICU mortality, hospital mortality, or hospital discharge as an ultimate outcome.

OTHER OUTCOMES:
Length of stay | Participants will be followed for the duration of hospital stay, an expected average of 6 days
  A secondary outcome of length of stay both in the Intensive Care Unit as well as total hospital stay after enrollment will be assessed.
Clinical Cure | Participants will be followed for the duration of hospital stay, an expected average of 6 days
  This secondary outcome measure is defined as resolution of sepsis. Clinical signs and symptoms present at the time of enrollment as well as the presence in any clinical cultures of antimicrobial resistant organisms not present prior to enrollment will be ascertained.

CONTACTS AND LOCATIONS:
Overall Officials: Ebbing Lautenbach, MD,MPH,MSCE, Principal Investigator — Univeristy of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania - Medical Intensive Care Unit, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No